CLINICAL TRIAL: NCT03872583
Title: Understanding Magnetic Resonance Imaging in Multiple Sclerosis - a Randomized, Controlled, Double Blind Trial
Brief Title: Understanding Magnetic Resonance Imaging in Multiple Sclerosis
Acronym: UMIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PV5722
Record Dates: First submitted 2019-01-25; First posted 2019-03-13 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Clinically Isolated Syndrome
Keywords: Patient education; Disease-specific knowledge; Shared decision making
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, physicians, outcome assessors and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Understanding MRI in MS (website) (Experimental): Participants will receive access to a newly developed, innovative, interactive and evidence-based education tool about magnetic resonance imaging in multiple sclerosis.
  Interventions: Other: Understanding MRI in MS (website)
- Control website (Active Comparator): Participants will receive access to a specifically designed control website containing the information about magnetic resonance imaging in multiple sclerosis, that is freely available on the websites of major European multiple sclerosis self help organization (Australia, Belgium, Canada, France, Germany, Great Britain, Netherland, USA).
  Interventions: Other: Control website

INTERVENTIONS:
Other: Understanding MRI in MS (website) — Access to an innovative, interactive and evidence-based online education tool about MRI in multiple sclerosis.
  Arms: Understanding MRI in MS (website)
Other: Control website — Access to a specifically designed control website containing information on MRI in MS freely available on the websites of major European MS self-help organizations.
  Arms: Control website

SUMMARY:
Magnetic resonance imaging (MRI) results play a major role in the lives of people with multiple sclerosis (pwMS). Even though MRI is used for diagnosis, prognosis and therapy control, pwMS' knowledge concerning this complex matter is scarce. Without adequate disease-specific knowledge, pwMS cannot truly make an informed choice when considering their MRI results (e.g. necessity of future MRI scans or therapy change).

The investigators have developed an innovative, evidence-based and interactive online education tool called "Understanding MRI in MS", which incorporates all relevant information about MRI in MS and its implications in disease management.

In this randomized, controlled and double-blind trial the tool's effect on MRI-specific knowledge, self-perceived competence and involvement in medical decision, that are based on MRI results will be assessed.

DETAILED DESCRIPTION:
For the randomized controlled trial (RCT), n=120 consecutive patients of 4 centers, for whom a brain (or brain and spine) MRI scan is planned within the next 6 months, will be invited to participate in the trial. Eligible patients will be asked to participate, and, if willing, will receive information about the study by the recruiting physician and written consent will be obtained. Participants will then answer a baseline questionnaire including demographic data, numeracy, attitude and emotions towards MRI (MRI-emotions and attitude questionnaire, MRI-EMA, newly developed) and MRI-specific knowledge (MRI-risk knowledge questionnaire 2.0, MRI-RIKNO 2.0, newly developed).

Patients will then be randomized into two groups: The intervention group of n=60 participants gets access to the web-based educational tool, the control group of n=60 to a sham intervention with standard information on MRI.

Participants will be asked to provide an e-mail address via which the login for the educational tool will be delivered. After two weeks participants will be asked to fill out the following tools:

Primary endpoint

* MRI-risk knowledge questionnaire 2.0 (MRI-RIKNO 2.0) (newly developed)
* MRI-emotions and attitude questionnaire (MRI-EMA) (newly developed)
* Threat by MS
* Autonomy preferences (Control Preference Scale)
* Subjective knowledge (VAS scale) (22)

Within the course of 2 weeks to 6 months the scheduled MRI will take place, followed by a patient-physician encounter, in which the MRI results are discussed. Directly after this encounter patients and physicians will be asked to answer MAPPIN'SDM questionnaires to assess perceived shared decision making behaviour and realization of autonomy preferences (Control reference scale). All patients will also be asked questions concerning any decisions taken based on the MRI, either a start/change of treatment or agreement on a new MRI in a defined time-frame. N=5 patients of each arm in the study center in Hamburg will be randomly selected and the communication of results during this consultation will be audiotaped and evaluated using the MAPPIN'SDM observer rating approach.

In a telephone follow-up after 6 months, implementation of the decisions will be checked.

ELIGIBILITY:
Inclusion Criteria:

* 18 years 65 years
* MRI within 6 weeks to 6 months
* internet access AND
* diagnosis of relapsing-remitting MS (RRMS) according to the McDonald criteria (Thompson et al., 2018), <10 years disease duration + active disease course (i.e. therapy change or new T2 lesion within the previous year) OR
* clinically isolated syndrome (CIS) (with at least one MS-typical T2 lesion)

Exclusion Criteria:

* diagnosis of secondary-progressive MS
* diagnosis of primary-progressive MS
* diagnosis or suspected central nervous system disease other than MS
* severe cognitive deficit
* major psychiatric illness
* patients who are related to medical personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging risk knowledge questionnaire 2.0 (MRI-RIKNO 2.0) | 2 weeks
  15-item magnetic resonance imaging-specific knowledge questionnaire (min. points 0, maximum points 22; higher values indicate greater knowledge)

SECONDARY OUTCOMES:
Emotions and attitude towards magnetic resonance imaging (MRI-EMA) | Baseline, 2 weeks
  Validated 10-item questionnaire on emotions and attitude towards magnetic resonance imaging, sub-scales (min. value: 1, max. value: 4; higher values indicate greater expression of the feature): 1) Fear of MRI scan, 2) Fear of MRI results, 3) Feeling of control, 4) Feeling of competence
Control preference scale (CPS) | Baseline, 2 weeks, after patient-physician encounter (i.e. 4 weeks to 6 months after baseline)
  Scale to assess autonomy preferences during medical decisions (5 categories between complete autonomy and paternalistic decision making as the extremes)
Threat by MS | baseline, 2 weeks
  Visual analogue scale to assess anxiety associated with disease progression (min. 0, max. 100; higher values indicate higher subjective threat)
Hospital Anxiety and Depression Scale (HADS) | Baseline, 2 weeks
  Questionnaire to assess anxiety and depression (min. 0, max. 42 points (21 points for each subscale, subscales are added); higher values indicate more severe depression/anxiety)
Multifocal Approach to Sharing in Shared Decision Making (MAPPIN'SDM) | after patient-physician-encounter (i.e. 4 weeks to 6 months after baseline)
  Tool to assess the amount of shared decision making during a patient-physician encounter (min. value 0, max. value 45; higher values indicated higher level of shared decision making)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, Prof., Principal Investigator — University Medical Center Hamburg-Eppendorf; Institute for Neuroimmunology and Multiple Sclerosis
Locations (1):
- University Medical Centre Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brand J, Kopke S, Kasper J, Rahn A, Backhus I, Poettgen J, Stellmann JP, Siemonsen S, Heesen C. Magnetic resonance imaging in multiple sclerosis--patients' experiences, information interests and responses to an education programme. PLoS One. 2014 Nov 21;9(11):e113252. doi: 10.1371/journal.pone.0113252. eCollection 2014. PMID 25415501
- [Background] Gaissmaier W, Giese H, Galesic M, Garcia-Retamero R, Kasper J, Kleiter I, Meuth SG, Kopke S, Heesen C. Numeracy of multiple sclerosis patients: A comparison of patients from the PERCEPT study to a German probabilistic sample. Patient Educ Couns. 2018 Jan;101(1):74-78. doi: 10.1016/j.pec.2017.07.018. Epub 2017 Jul 17. PMID 28764895
- [Background] Heesen C, Kasper J, Fischer K, Kopke S, Rahn A, Backhus I, Poettgen J, Vahter L, Drulovic J, Van Nunen A, Beckmann Y, Liethmann K, Giordano A, Fulcher G, Solari A; AutoMS-group. Risk Knowledge in Relapsing Multiple Sclerosis (RIKNO 1.0)--Development of an Outcome Instrument for Educational Interventions. PLoS One. 2015 Oct 2;10(10):e0138364. doi: 10.1371/journal.pone.0138364. eCollection 2015. PMID 26430887
- [Background] Heesen C, Kasper J, Kopke S, Richter T, Segal J, Muhlhauser I. Informed shared decision making in multiple sclerosis--inevitable or impossible? J Neurol Sci. 2007 Aug 15;259(1-2):109-17. doi: 10.1016/j.jns.2006.05.074. Epub 2007 Apr 2. PMID 17400253
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Boeije HR, Janssens AC. 'It might happen or it might not': how patients with multiple sclerosis explain their perception of prognostic risk. Soc Sci Med. 2004 Aug;59(4):861-8. doi: 10.1016/j.socscimed.2003.11.040. PMID 15177841
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Riechel C, Alegiani AC, Kopke S, Kasper J, Rosenkranz M, Thomalla G, Heesen C. Subjective and objective knowledge and decisional role preferences in cerebrovascular patients compared to controls. Patient Prefer Adherence. 2016 Aug 2;10:1453-60. doi: 10.2147/PPA.S98342. eCollection 2016. PMID 27536077
- [Background] Kasper J, Hoffmann F, Heesen C, Kopke S, Geiger F. MAPPIN'SDM--the multifocal approach to sharing in shared decision making. PLoS One. 2012;7(4):e34849. doi: 10.1371/journal.pone.0034849. Epub 2012 Apr 13. PMID 22514677
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Schiffmann I, Freund M, Vettorazzi E, Stellmann JP, Heyer-Borchelt S, D'Hooghe M, Haussler V, Rahn AC, Heesen C. Assessing the effect of an evidence-based patient online educational tool for people with multiple sclerosis called UMIMS-understanding magnetic resonance imaging in multiple sclerosis: study protocol for a double-blind, randomized controlled trial. Trials. 2020 Dec 9;21(1):1008. doi: 10.1186/s13063-020-04855-5. PMID 33298133

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03872583/SAP_000.pdf